CLINICAL TRIAL: NCT06310057
Title: Tofacitinib in the Treatment of Refractory Axial Spondyloarthritis Patients: A Dose Escalation Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh (Other)
Collaborators: Incepta Pharmaceuticals Ltd (Industry)
Responsible Party: Principal Investigator, Abdul Mahin Tazbir, MD Resident, Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4139
Record Dates: First submitted 2024-03-08; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Axial Spondyloarthritis
MeSH Terms: conditions — Axial Spondyloarthritis | interventions — tofacitinib

STUDY DESIGN:
Intervention Model Description: Dose escalation study, all the patients will recieve 10mg tofacitinib at the beginning. Then at 3rd month, one group will continue at 10mg, if they fulfill the ASDAS major improvement criteria and other group will escalate to 15mg.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tofacitinib 10mg (Experimental): All patient that fulfill the inclusion ans exclusion criteria will start at 10mg tofacitinib.
  Interventions: Drug: Tofacitinib
- Tofacitinib 15 mg (Experimental): At 3rd month, patients that do not fulfill the ASDAS major improvement criteria will get 15mg tofacitinib.
  Interventions: Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib (JAKi) is a targeted therapy option for patients with refractory ax-SpA.

SUMMARY:
The goal of this clinical trial is to assess the efficacy of tofacitinib in refractory axial spodyloarthritis (ax-SpA) with dose escalation from 10mg to 15mg. Patients will start on 10mg and then divided into 2 groups (10 and 15) at 3rd month according to major improvement criteria.

The main question[s] it aims to answer are:

* Efficacy and safety of tofacitinib in different doses
* If escalation of tofacitinib is justified if clinical criteria is not fulfilled at 10mg

DETAILED DESCRIPTION:
Axial spondyloarthritis (ax-SpA) is a major cause of chronic low back pain in the young. It causes significant disability and impairs quality of life. Management of (ax-SpA) includes physical therapy along with NSAIDs, followed by TNFi or IL-17i or JAKi in refractory ax-SpA. In Bangladesh, TNFi and IL-17i are expensive, whereas Tofacitinib (JAKi) is affordable and widely used in Bangladesh. However, recent study shows that a significant number of patients, 39.4% do not meet criteria for ASDAS CRP clinically important criteria and only 26% meets the criteria for ASDAS major improvement to tofacitinib 10mg daily. 102 patients of refractory ax-SpA meeting the enrollment criteria will be taken and put on 10mg tofacitinib. Those who fail to attain ASDAS CRP major improvement criteria at 12 weeks will be put on 15mg tofacitinib and both the groups will be compared at week 24 in a dose escalation study.

No studies have been done on 15mg tofacitinib for ax-SpA, such a study will provide us ground for escalation of tofacitinib. Regarding safety issues, FDA has warned against the use of 20mg tofacitinib but not for 15mg. Baseline characteristics and variables will be recorded at initiation of therapy, 4th, 12th and 24th week. The study will take place in Rheumatology outdoor, BSMMU and Modern One Stop Arthritis Care and Research Centre, Dhaka from July 2022- April 2024. Patient's socio-demographic and clinical data will be taken in a semi-structured questionnaire. At every follow up detailed history, thorough physical examination and investigations will be done to evaluate the efficacy and adverse effects. Patients will be assessed for response, ASDAS-CRP, ASDAS-ESR, ASAS-20, BASFI, BASDAI, BASMI, ASQoL, SF-36, MASES and VAS will be noted. CBC, CRP, S. creatinine and S. ALT will be done during follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Patient fulfill the ASAS classification criteria for ax-SpA
3. Patient fulfill the definition of refractory axial ax-SpA
4. Patients with ASDAS-CRP>2.1

Exclusion Criteria:

1. Patient currently taking or had prior treatment with bDMARD or tsDMARD (including JAK inhibitor)
2. Patient with any active or history of any chronic or recurrent or serious or opportunistic infection/sepsis (including tuberculosis)
3. Hemoglobin (Hb) < 9 g/dl
4. White blood cell count < 4000, Neutrophil count < 1000, Platelet count < 100000/mm3
5. Live vaccines within 3 months prior to the first dose
6. GFR less than 50 mL/min
7. Alanine aminotransaminase (ALT) more than 2 times of ULN
8. Pregnant or breast feeding females of child-bearing potential not using highly effective contraception
9. Evidence or history of malignancy
10. New York Heart Association Class III and IV congestive heart failure
11. Any lymphoproliferative disorder, history of lymphoma, leukemia, or signs and symptoms suggestive of current lymphatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
To assess the ASDAS CRP major improvement criteria in refractory ax-SpA patients with dose escalation from 10mg to 15mg | 6 months
  To assess the ASDAS CRP major improvement criteria in refractory ax-SpA patients with dose escalation from 10mg to 15mg

SECONDARY OUTCOMES:
Clinicodemographic characteristics of Ax-SpA, ASDAS CRP outcome rates, quality of life, adverse effects | 6 months
  1. To compare the clinicodemographic characteristics of refractory ax-SpA patients with and without ASDAS CRP major improvement outcome
  2. To determine the ASDAS CRP outcome rates with 10 mg and 15mg tofacitinib
  3. To evaluate the change in quality of life with the outcome of ASDAS CRP
  4. To evaluate the adverse effects of 10 mg and 15 mg tofacitinib

CONTACTS AND LOCATIONS:
Locations (1):
- Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh